CLINICAL TRIAL: NCT02524405
Title: The Brain Eye Amyloid Memory (BEAM) Study: Validation of Ocular Measures as Potential Biomarkers for Early Detection of Brain Amyloid and Neurodegeneration
Brief Title: BEAM: Brain-Eye Amyloid Memory Study
Acronym: BEAM
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Brain Canada (Other); Weston Brain Institute (Other); GE Healthcare (Industry); University Health Network, Toronto (Other); Centre for Addiction and Mental Health (Other); Baycrest (Other); Unity Health Toronto (Other); Kensington Eye Institute (Other)
Responsible Party: Principal Investigator, Dr. Sandra E Black, Principal Investigator, Sunnybrook Health Sciences Centre
Other Study IDs: 221-2013
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment; Vascular Cognitive Impairment; Parkinson's Disease; Lewy Body Disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Parkinson Disease; Lewy Body Disease | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples for genetic testing including apoliprotein E4 status, as well as for proteomic, lipidomic and other fluid biomarkers of neurodegeneration and vascular disease, will be collected for each participant. All samples should be taken after a 10 hour fast; if not possible, the participant should have a light meal only. Samples should be collected between 8am and 10am, in order to minimize circadian variations in biomarker levels.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Normal Controls: Upto 85 normal elders, 50-90 years old who are within normal limits on the study neuropsychological battery will be enrolled. All patients involved in the study will undergo SD-OCT, eye tracking, gait and balance assessments, blood draw for genomics and fluid biomarkers, neuropsychological assessment, brain MRI and brain amyloid PET.
  Interventions: Other: Pittsburgh Compound B [11C]-PIB
- Alzheimer's Disease (AD): Sixty-five subjects meeting the National Institute on Aging-Alzheimer's Association (NIA-AA) core clinical criteria for probable AD dementia will be enrolled. All patients will undergo SD-OCT, eye tracking, gait and balance assessments, blood draw for genomics and fluid biomarkers, neuropsychological assessment, brain MRI and brain amyloid PET. A subset will undergo SV-OCT.
  Interventions: Other: Pittsburgh Compound B [11C]-PIB
- Mild Cognitive Impairment (VCI): Sixty-five subjects meeting the National Institute on Aging-Alzheimer's Association criteria for amnestic or multi-domain MCI with MoCA score ≥18 will be enrolled. All patients will undergo SD-OCT, eye tracking, gait and balance assessments, blood draw for genomics and fluid biomarkers, neuropsychological assessment, brain MRI and brain amyloid PET. A subset will undergo SV-OCT.
  Interventions: Other: Pittsburgh Compound B [11C]-PIB
- Subcortical Vascular Impairment (VCI): Sixty-five subjects meeting the American Heart Association-American Stroke Association (AHA-ASA) criteria for probable vascular dementia (VaD) or probable vascular mild cognitive impairment (VaMCI) due to subcortical ischemic vascular disease , and probable or possible Cerebral Amyloid Angiopathy using the Modified Boston Criteria116 will be enrolled. All patients will undergo SD-OCT, eye tracking, gait and balance assessments, blood draw for genomics and fluid biomarkers, neuropsychological assessment, brain MRI and brain amyloid PET. A subset will undergo SV-OCT.
  Interventions: Other: Pittsburgh Compound B [11C]-PIB
- LBD Spectrum: Sixty- five subjects with: Dementia with Lewy Bodies (DLB) meeting the criteria for probable Dementia with Lewy Bodies with MMSE score ≥20; or PD-MCI meeting the proposed Level I criteria for Mild Cognitive Impairment in Parkinson's Disease with MoCA score 18-24; or; PDD meeting the criteria for probable Parkinson's Disease - Dementia and MMSE score ≥20 will be enrolled. All patients involved will undergo SD-OCT, eye tracking, gait and balance assessments, blood draw for genomics and fluid biomarkers, neuropsychological assessment, brain MRI and brain amyloid PET. A subset will undergo SV-OCT.
  Interventions: Other: Pittsburgh Compound B [11C]-PIB

INTERVENTIONS:
Other: Pittsburgh Compound B [11C]-PIB — This is a cross-sectional study of patients with various forms of cognitive impairment and a healthy control group for comparison. Brain amyloid PET scans using the radioligand Pittsburgh Compound B [11C]-PIB, which is not yet approved for clinical use in Canada, will be performed in all subjects.

SUMMARY:
The main objectives for this study are:

1. To investigate novel, non-invasive ocular measurements including optical coherence tomography and eye tracking in a cross-sectional study of participants with various neurodegenerative dementias against standard cognitive assessments and brain imaging measures; and
2. To assess the potential utility of ocular assessments for early detection in the pre-dementia, i.e. the so-called Mild Cognitive Impairment (MCI) stage, across the common neurodegenerative dementia syndromes and, Vascular Cognitive Impairment (VCI) due to small vessel disease (SVD).
3. To determine the prevalence and relevance of amyloid uptake on PET scanning across the dementias most commonly associated with amyloidosis. Specifically we aim to examine correlations with amyloid uptake status in patients symptomatic from the most common proteinopathies (ie amyloid, tau, synuclein) combined in varying degrees with the most common vasculopathies (ie small vessel disease) using multimodal structural and functional imaging, cognitive behavioral, and gait and balance measures, taking into account genetic risk markers (particularly apolipoprotein E genotypes) and fluid biomarkers ( eg cytokines, oxidative stress, lipidomics).

DETAILED DESCRIPTION:
1. Retinal correlations with neurodegeneration:

   1. Retinal nerve fiber layer (RNFL) pattern will differ in participants in the MCI and early stages of LBD spectrum, AD, and VCI, relative to normal elders. i) RNFL thinning around the optic disc and macular thinning will correlate with hippocampal atrophy and with the cortical thickness signature of MCI and AD2-4. ii) If detected in the other disorders, RNFL thinning will also correlate with this topographical AD pattern of atrophy in those who are amyloid positive on PET. iii) Retinal and cortical thinning will predict brain amyloid PET. iv) Selective peripapillary RNFL thinning in the superior and inferior quadrants described in MCI/milder AD cases will correlate with precuneus and lingual gyrus cortical thinning respectively.
   2. Retinal artery narrowing will correlate with presence of covert lacunar infarcts and retinal venular widening with moderate to severe periventricular white matter hyperintensities.
2. Amyloid deposition above accepted cut-offs will vary across the 4 cohorts and when present will correlate meaningfully with cognitive and behavioural patterns, including ocular (retinal and eye tracking), gait and balance measures and brain imaging results.

Specific hypotheses are:

1. Apoelipoprotein E e4 carrier status will increase likelihood of amyloid positivity across the cohorts.
2. Amyloid positivity will be associated with poorer short term memory performance, smaller hippocampal volumes, greater cortical thinning in signature areas traditionally associated with Alzheimer's disease, and also with lobar microbleed counts.
3. Small Vessel Disease burden as quantified on PD/T2 and FLAIR MRI will be associated with speed of processing, attention and executive functions and with a different pattern of cortical thinning involving more inferior and medial frontal regions.
4. Amyloid deposition as measured by regional standardized uptake value ratio (SUVR), and Small Vessel Disease burden will correlate differentially with structural imaging measures, as well as both functional and structural brain connectivity measures.

Study Procedures Overview The study procedures are listed below in the recommended order of assessment but may be performed in any sequence (with specific exceptions as described). Multiple assessments may be performed on the same day for participant convenience. Brain imaging and neuropsychology procedures should be completed within 4 months of screening.

Screening Visit Consent. The study will be explained and written informed consent for participation will be obtained from the patient or his/her substitute decision maker and the participant's study partner (if applicable).

Screening. The general and disease-specific inclusion and exclusion criteria will be assessed. If the MMSE, MoCA, DOC (Depression, Obstructive Sleep Apnea, Cognition) questionnaire and/or TorCA (formally known as Behavioural Neurology Assessment - Revised (BNA-R) have not been administered within the past four months, they will be administered at the screening visit. Information on the patient's concomitant medications, medical, surgical, ophthalmological history, family health history and other relevant history will be collected, as well as information on both the patient's and the study partner's demographics. The patient's corrected near visual acuity will be checked. Auditory acuity at various frequencies will be assessed using an audiometer. Fasting blood will be drawn, for analysis of HbA1c, CBC, electrolytes, creatinine, urea, lipid profile, glucose, liver function (AST, ALT, ALP, bilirubin), homocysteine, B12 and TSH. Blood will also be drawn for genomics and fluid biomarkers (see next section.)

Genomics and Fluid Biomarkers. Fasting blood samples for genetic testing including apoliprotein E4 status, as well as for proteomic, lipidomic and other fluid biomarkers of neurodegeneration and vascular disease, will be collected from each participant.

Neuropsychological Battery and Questionnaires. The cognitive battery comprises most of the tests used in the Ontario Neurodegenerative Disease Research Initiative (ONDRI) study, a new province-wide neurodegeneration research collaboration, with some modifications. It includes measures of executive function, memory, language, and visuospatial ability. Function, mood and behaviour, and caregiver burden will also be assessed using the questionnaires used in ONDRI. The full list of the assessment procedures is included in the BEAM neuropsychology manuals.

SD-OCT. Assessments to meet ocular criteria will include visual acuity, intra-ocular pressure (IOP) measurement and a non-mydriatic fundus camera recording, performed by a certified ophthalmic technician. The participant will then undergo SD-OCT to determine retinal nerve fiber layer thickness.

Vital Signs and Neurological Exam. Vital signs will be measured and a neurological examination will be performed.

Gait and Balance Assessment. Information on aid use and balance will be collected using questionnaires. Participants' leg length, calf circumference, height, and weight will be measured and recorded when possible.

Eye Tracking. Participants will be asked to look at a computer monitor and perform three sets of tasks (pro-saccade, anti-saccade, and dynamic free viewing) while a specialized camera tracks and records their eye movements. Participants who are unable to complete these assessments will be allowed to continue participation in the study.

SV-OCT at Sunnybrook. SV-OCT will be done in subsamples with high SVD vs. minimal SVD loads. A rapid (>100 fps) 3D scanning protocol will be applied to SD-OCT, allowing acquisition of speckle variance due to microscopic blood flow in the retinal vasculature. Image processing using GPU based technique will provide real-time assessment of microvasculature morphology.

MRI. 3DT1 SPGR, interleaved spin echo PD/T2 and FLAIR to assess SVD, and gradient echo images to assess microbleeds, will be obtained on the 3 Tesla scanners at each of the TDRA sites. The PD/T2 and FLAIR images are co-registered to the T1-weighted image to remove non-brain tissues to determine total supratentorial intracranial volume to correct for head size, classify brain tissue compartments and automatically identify subcortical and white matter hyperintensities using a published in-house pipeline, "Lesion Explorer", which with manual editing yields number, size, location, and volume of the hyperintensities. For hippocampal volume, we use our fully automated segmentation pipeline based on a template library registration117, 118. We will also acquire DTI to generate total and regional fractional anisotropy (FA) and Mean Diffusivity Maps, using FSL and DTI tool box, and a resting state fMRI to explore Default Mode Network (DMN) connectivity, using a processing pipeline steps previously applied to AD patients and controls119.

Arterial Spin Labeling (ASL) will be included at certain sites which are capable of acquiring this sequence, to obtain measures of regional cerebral perfusion.

Amyloid PET. PIB, labelled with the positron emitting atom carbon-11, is a radiotracer that targets Aβ-aggregates (β-amyloid) in vivo. β-amyloid deposits are present in the brain of patients with Alzheimer's Disease (AD). Therefore, Aβ-plaques in the brain may be a useful biomarker of the disease and its progression and [11 C]-PIB may be a useful tool to detect these plaques in the human living brain with PET.

[11 C ]-PIB is an investigational positron emitting radiopharmaceutical (PER) not yet marketed in Canada. The ligand will be manufactured at CAMH PET centre. PET imaging will be performed using [11 C] PIB at CAMH PET Centre with PET/CT-Discovery MI scanner using the standardized acquisition protocol.

The PET imaging protocol begins with a low dose CT scan (less than 0.05 mSv) for attenuation correction. Immediately following this acquisition, a bolus containing approximately 10 ± 1 mCi of [11 C]-PIB is administered by IV injection, followed by 90 minutes acquisition. Acquisition and reconstruction of PET images are done according to the standard PET Centre Imaging Protocols.

Phone Check Ups: For safety measures the participants will be contacted by phone to discuss any possible adverse event and general well-being two times during the course of the study:

* 24-72 hours after the PET scan
* 30 days (+/- 7 days) after PET Scan and/or the last study procedure

ELIGIBILITY:
General Inclusion Criteria (All Subgroups)

Participants must meet each of the following criteria for enrolment into the study:

1. Written informed consent obtained and documented
2. Male or post-menopausal female (minimum of one year since the last menstrual period)
3. 50-90 years of age
4. Self-reported proficiency in speaking and understanding spoken English questions
5. ≥8 years education
6. Capable of cooperating for the duration of the study procedures and assessments
7. Willing to undergo study procedures and remain unaware of the results (unless there are findings that are of clinical significance and would require further action, in the opinion of the study physician)
8. Sufficient vision to participate in cognitive testing (corrected near visual acuity of Snellen 20/70 in at least one eye) and eye-tracking (able to identify symbols and stimuli presented on a computer screen in front of them)
9. Sufficient corrected hearing to participate in cognitive testing
10. Good venous access for phlebotomy to be performed
11. Able to walk, with or without an assistive aid (e.g., cane, walker)

Subgroup-Specific Inclusion Criteria

Cognitively Normal Controls

1. Cognitively normal and functionally independent in pre-screening history
2. Within normal limits on the TorCA (formally known as Behavioural Neurology Assessment - Revised (BNA-R)
3. Within normal limits on the study neuropsychological battery

Mild Cognitive Impairment (MCI)

1. Meets the National Institute on Aging-Alzheimer's Association criteria for single or multi-domain amnestic MCI
2. Impairment of episodic memory plus or minus other cognitive domains on the TorCA
3. Montreal Cognitive Assessment (MoCA) score ≥18
4. Mini-Mental State Examination (MMSE) > 20
5. In the opinion of the investigator if required: reliable and capable partner who has regular interaction with them, can provide a collateral history, can assist in compliance with study procedures, and who is willing to act as the Study Partner (provide written informed consent) and remain unaware of the results

Alzheimer's Disease (AD)

1. Meets the National Institute on Aging-Alzheimer's Association (NIA-AA) core clinical criteria for probable or possible AD dementia
2. Mild early AD stage, as defined by MMSE score ≥18, Atypical cases with a MoCA ≥ 14 will also be allowed.
3. Impairment in two or more cognitive domains on the TorCA
4. Reliable and capable partner who has regular interaction with them, can provide a collateral history, can assist in compliance with study procedures, and who is willing to act as the Study Partner (provide written informed consent) and remain unaware of the results

Lewy Body Disease (LBD) Spectrum PD-MCI

1. Meets the proposed Level I criteria for Mild Cognitive Impairment in Parkinson's Disease
2. MMSE score ≥20
3. MoCA score ≥18
4. Hoehn & Yahr stage 1-3
5. Reliable and capable partner who has regular interaction with them, can provide a collateral history, can assist in compliance with study procedures, and who is willing to act as the Study Partner (provide written informed consent) and remain unaware of the results

LBD-MCI

1. Meets the criteria for Dementia with Lewy Bodies (McKeith et al, 2017 in press)but has preserved daily functioning
2. MMSE score ≥20
3. MoCA score ≥18
4. Hoehn & Yahr stage ≤3
5. Reliable and capable partner who has regular interaction with them, can provide a collateral history, can assist in compliance with study procedures, and who is willing to act as the Study Partner (provide written informed consent) and remain unaware of the results

Dementia with Lewy Bodies (DLB)

1. Meets the criteria for probable or possible Dementia with Lewy Bodies (McKeith et al, 2017 in press)
2. MMSE score ≥14
3. MoCA score ≤25
4. Reliable and capable partner who has regular interaction with them, can provide a collateral history, can assist in compliance with study procedures, and who is willing to act as the Study Partner (provide written informed consent) and remain unaware of the results

PDD

1. Meets the criteria for probable Parkinson's Disease - Dementia
2. MMSE score ≥18
3. MoCA score ≤25
4. Hoehn & Yahr stage ≤4
5. Reliable and capable partner who has regular interaction with them, can provide a collateral history, can assist in compliance with study procedures, and who is willing to act as the Study Partner (provide written informed consent) and remain unaware of the results

Subcortical Vascular Cognitive Impairment (VCI)

1. Presence of subcortical vascular disease, indicated by the following:

   i. Periventricular Fazekas score = 3, with or without subcortical lacunes or small cortical infarcts (<1.5 cm in longest diameter); or ii. Fazekas score ≥ 2, with 2 or more subcortical lacunes or small cortical infarcts (<1.5 cm in longest diameter); or iii. Fazekas score = 0 or 1, with 3 subcortical lacunar infarcts (<1.5 cm in diameter), at least 1 in each hemisphere; or

   iv. Probable or possible Cerebral Amyloid Angiopathy using the Modified Boston Criteria
2. Reliable and capable partner who has regular interaction with them, can provide a collateral history, can assist in compliance with study procedures, and who is willing to act as the Study Partner (provide written informed consent) and remain unaware of the results

Exclusion criteria General Exclusion Criteria (All Subgroups)

Participants who exhibit any of the following conditions will be excluded from the study:

1. Underlying conditions (other than the disease being studied) which in the opinion of the investigator may interfere with the participant's ability to participate in the study or may compromise study results, including but not limited to:

   1. Unstable cardiac, pulmonary, renal, hepatic, endocrine (i.e. diabetes) or hematologic disease
   2. Active malignancy or infectious disease
   3. Significant psychiatric illness, including life-long depressive illness
   4. History of significant learning disability
   5. Significant other neurologic disease (e.g., multiple sclerosis, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma) or cognitive complications of cancer
   6. Symptomatic stroke within the past 6 months
   7. Substance abuse within the past year or history of alcohol or drug abuse which in the opinion of the investigator may interfere with the participant's ability to comply with the study procedures
   8. History of significant head trauma or recurrent concussions requiring hospitalization followed by persistent neurologic defaults or known structural brain abnormalities
   9. Pain or sleep disorder that could interfere with cognitive testing
   10. Any disability that would limit the ability to perform study assessments
2. Ocular conditions, including:

   a. Clinical diagnosis of glaucoma, taking eye drops for glaucoma, or previous surgery (including laser) for glaucoma b. Any other serious eye disease or treatment or eye surgery, including any history of intra-vitreal injections c. History of optic neuritis d. Previous retinal laser therapy (either pan-retinal, or grid/focal) for diabetic retinopathy e. Cupping of the optic nerve head (ONH) consistent with a diagnosis of glaucoma, as clinically determined by expert ophthalmological assessment of digital colour fundus images centered on the ONH. Specifically, one or more of the following (assessed as part of SD-OCT visit at Kensington Eye Institute): i. a cup/disc ratio of 0.7 or greater in either eye ii. a cup/disc asymmetry of more than 0.2 iii. disc hemorrhage iv. notch f. Wet/exudative age-related macular degeneration (ARMD) in one or both eyes, as clinically determined by expert ophthalmological assessment of digital color fundus images centered on the fovea (assessed as part of SD-OCT visit at Kensington Eye Institute)
3. Intra-ocular pressure greater than 22mmHg or a difference in intra-ocular pressure (Goldmann tonometry) greater than 5mmHg between the two eyes (assessed as part of SD-OCT visit at Kensington Eye Institute)
4. Brain imaging abnormalities detected either on clinical MRI or CT prior to enrollment or on study MRI, including but not limited to:

   1. Evidence of infection
   2. Focal compressive mass lesions (tumours, subdural hematomas, malformations, etc.)
5. Known hypersensitivity to Pittsburgh Compound B [11C]-PIB or any components of the[11C]-PIB Injection formulation
6. Contraindications to 3T MRI, as listed in the site-specific Magnetic Resonance Environment Screening Questionnaire (e.g. metal implant)
7. Unable to tolerate the MRI environment (e.g., due to physical size and/or claustrophobia)
8. Currently enrolled in a disease-modifying therapeutic trial that in the opinion of the Principal Investigator can potentially compromise study results

Subgroup-Specific Exclusion Criteria Cognitively Normal Controls

1. Subjective memory complaints
2. Brain imaging abnormalities detected either on clinical MRI or CT prior to enrollment or on study MRI, including but not limited to:

   1. Periventricular Fazekas score = 2.5 or 3
   2. Subcortical non-lacunar infarct or more than 1 subcortical lacunar infarct (<1.5 cm in longest diameter)
   3. Cortical ischemic stroke Cortical or subcortical hemorrhagic stroke >1.5cm in diameter

MCI, AD, and LBD Spectrum

(1) Brain imaging abnormalities detected either on clinical MRI or CT prior to enrollment or on study MRI, including but not limited to:

1. Periventricular Fazekas score = 2.5 or 3
2. Subcortical non-lacunar infarct or more than 1 subcortical lacunar infarct (<1.5 cm diameter)
3. Cortical ischemic stroke >1.5cm in longest diameter
4. Cortical or subcortical hemorrhagic stroke >1.5cm in diameter

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three hundred and forty five (345) participants will be enrolled: upto 85 cognitively normal elders, 65 with MCI, 65 with AD, 65 with LBD spectrum disease, and 65 with subcortical Vascular Cognitive Impairment.
  All patients will receive a standardized work up for dementia including brain imaging and a blood work screen to rule out secondary causes of dementia as part of their clinical work-up prior to study enrollment. Memory clinic patients will undergo a detailed neurocognitive assessment (Toronto Cognitive Assessment - TorCA), and the clinical history and examination will use a standardized common elements approach.
Sampling Method: Non-Probability Sample
Enrollment: 345 (Estimated)
Dates: Start 2016-02; Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Retinal nerve fiber layer thickness | One-time assessment
  This potential ocular biomarker will compared among the different cohorts and be validated against brain MRI and brain amyloid PET.
Amyloid Depostition | One-time assessment
  This will be compared among the different cohorts and be validated against brain amyloid PET, and are expected to correlate meaningfully with cognitive and behavioural patterns, including retinal and eye-tracking, gait and balance.

SECONDARY OUTCOMES:
Retinal artery narrowing | One-time assessment
  The extent of correlation between retinal artery narrowing and the presence of covert lacunar infarcts on MRI will be assessed.
Retinal venular widening | One-time assessment
  The extent of correlation between retinal venular widening and the amount of periventricular white matter hyperintensities on MRI will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Black, MD, Principal Investigator — Sunnybrook Health Sciences Center
Locations (5):
- Canada (5):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Baycrest Health Sciences, Toronto, Ontario
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario